CLINICAL TRIAL: NCT03220490
Title: Efficacy and Necessity of Time Interval Between Instillation of Two Glaucoma Eye Drops
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-17-3820-AL-CTIL
Record Dates: First submitted 2017-06-19; First posted 2017-07-18 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Glaucoma; Glaucoma; Drugs
MeSH Terms: conditions — Glaucoma | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Short term: interval no-interval eye (Experimental): On the first day of the study, in the selected eye the investigators will examine the short term effect of IOP reduction of Brimonidine and Timolol with time interval.
  One drop of two types of IOP reduction drugs (Brimonidine and Timolol) will be given with a 5 minutes interval between the first (Brimonidine) and the second (Timolol) drop. IOP measurements will be taken every hour up to 6 hours after treatment.
  On the second day of the study (two weeks after the first day) the investigators will examine the short term effect of IOP reduction of Brimonidine and Timolol no time interval. Again one drop of the same two types of drugs will be given at the same order but with no time interval between them. IOP measurements will be taken in the same manner as on the first day.
  Interventions: Drug: IOP reduction of Brimonidine and Timolol with time interval; Drug: IOP reduction of Brimonidine and Timolol no time interval
- Short term: No-interval interval eye (Experimental): On the first day of the study, in the selected eye the investigators will examine the short term effect of IOP reduction of Brimonidine and Timolol with time interval.
  One drop of two types of IOP reduction drugs (Brimonidine and Timolol) will be given with no waiting period between the first (Brimonidine) and the second (Timolol) drop. IOP measurements will be taken every hour up to 6 hours after treatment.
  On the second day of the study (two weeks after the first day) the investigators will examine the short term effect of IOP reduction of Brimonidine and Timolol with time interval. Again one drop of the same two drugs will be given at the same order but with a five minute time interval between the first and second drop. IOP measurements will be taken in the same manner.
  Interventions: Drug: IOP reduction of Brimonidine and Timolol with time interval; Drug: IOP reduction of Brimonidine and Timolol no time interval
- Long term: interval no-interval eye (Experimental): In the first phase the effect of 5 minute interval between regular glaucoma drops - long term will be examined. The patients will be asked in this eye to wait 5 minutes after taking one of their IOP reduction drugs, before instilling the second type for a total duration of 1 month.
  After the one month has passed IOP measurement will be taken and the patients will be asked to switch to the no interval between regular glaucoma drops - long term phase in which they will be asked to take the drops for this eye at the same order but with no waiting period for a duration of 1 month. After the second month has passed IOP measurements will be repeated.
  Interventions: Behavioral: 5 minute interval between regular glaucoma drops - Long term; Behavioral: no interval between regular glaucoma drops - Long term
- Long term: No-interval interval eye (Experimental): In the first phase no interval between regular glaucoma drops - Long term will be examined. The patients will be asked in this eye to take both IOP reduction drugs, with no waiting period between them for a total duration of 1 month.
  After the one month has passed IOP measurement will be taken and the patient will be asked to switch to the to 5 minute interval between regular glaucoma drops - Long term phase and take the drops for the same eye at the same order but with a five minute waiting period for a duration of 1 month. After the second month has passed IOP measurements will be repeated.
  Interventions: Behavioral: 5 minute interval between regular glaucoma drops - Long term; Behavioral: no interval between regular glaucoma drops - Long term

INTERVENTIONS:
Behavioral: 5 minute interval between regular glaucoma drops - Long term — In the selected eye, the patient will be asked to take his two regular IOP reduction drugs while keeping a five minute time interval between instillation of the first and second drug for a duration of one month.
  Other Names: Long - interval
  Arms: Long term: No-interval interval eye; Long term: interval no-interval eye
Behavioral: no interval between regular glaucoma drops - Long term — In the selected eye, the patient will be asked to take his two regular IOP reduction drugs one after the other with no waiting period for a duration of one month.
  Other Names: Long - no interval
  Arms: Long term: No-interval interval eye; Long term: interval no-interval eye
Drug: IOP reduction of Brimonidine and Timolol with time interval — In the selected eye the subject will be given two types of IOP reduction drops: first "Brimonidine", "Alphagan®" (an alpha-agonist) followed by "Timolol", "Tiloptic®" (a beta-blocker). The drops will be given with a time interval of five minutes between the first and second drop.
  Other Names: Short - interval
  Arms: Short term: No-interval interval eye; Short term: interval no-interval eye
Drug: IOP reduction of Brimonidine and Timolol no time interval — In the selected eye the subject will be given two types of IOP reduction drops:first "Brimonidine", "Alphagan®" (an alpha-agonist) followed by "Timolol", "Tiloptic®" (a beta-blocker). The drops will be given one after the other with no waiting period.
  Other Names: Short - no interval
  Arms: Short term: No-interval interval eye; Short term: interval no-interval eye

SUMMARY:
According to the American Academy of Ophthalmology's Preferred Practice Pattern on Primary Open Angle Glaucoma, patients should wait five minutes between administering topical drops for intra-ocular pressure reduction.

To date, no study has shown the efficacy of this waiting period. In this study, we aim to establish the clinical significance of keeping a time interval between glaucoma medications.

DETAILED DESCRIPTION:
Glaucoma is a chronic disease in which constant damage to retinal nerve fibers. In most cases the damage is caused by increased intra-ocular pressure (IOP). Without treatment, this disease can cause irreversible decrease in visual fields until the patient eventually becomes blind.

The first line of treatment include topical eye-drops aimed at reducing IOP. Many patients require more than one drug type.

According to the American Academy of Ophthalmology's Preferred Practice Pattern on Primary Open Angle Glaucoma, patients who are using two or more drop types, should wait five minutes after the first drop, before administering the second type..

To date, no study has shown the efficacy of this waiting period. In this study, we aim to establish the clinical significance of keeping a time interval between glaucoma medications.

The study composes of two separate parts:

Part 1 - The aim of this part will be to estimate the short term effect on IOP reduction. Healthy subjects willing to participate voluntarily, will be given two IOP reduction drugs (Tilopitc and Alphagan) at different intervals in each eye. After which they will undergo repeated IOP measurements over a course of 7 hours.

Part 2 - The aim of this part will be to estimate the short term effect on IOP reduction. Glaucoma patients treated in the glaucoma clinic at Sheba-Medical center who are taking two different types of IOP reduction drugs in both eyes, will be recruited. The patients will be asked to keep a constant 5 minute interval between drops in one eye and to instill the drops in the other eye with no waiting time. After one month the patients will return for a revaluation of IOP and then be asked to switch the eyes so that the eye in which the interval was not kept will now be the one in which the drop will be put after 5 minute interval.

ELIGIBILITY:
Inclusion Criteria:

Short duration group

* Healthy individuals with negative past ocular history
* able to give consent

Long duration group:

* Diagnosed with primary open angle glaucoma and being treated with two types of IOP reduction drops.
* No other medical ocular history.
* No cognitive disfunction
* able to give consent
* No known arrhythmia

Exclusion Criteria (Both groups):

* Corneal disease preventing from visualization of the angle
* Closed angle
* Pregnant women
* Previous ocular surgery (including cataract or refractive surgery)
* Known allergy to ocular drops used in this study (e.g. brimonidine, timolol)
* History of asthma or arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Acute group - difference in IOP reduction | Six hour after taking the drops
  Difference in IOP change from baseline between the two eyes after treatment
Chronic group - change in IOP | one month
  Difference between eye in IOP change from baseline after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No